CLINICAL TRIAL: NCT04701983
Title: Randomized, Double-blind, Placebo-controlled, Parallel Group Phase 3 Study to Evaluate the Efficacy, Safety, and Tolerability of SAR440340/REGN3500/Itepekimab (Anti-IL-33 mAb) in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Study to Assess the Efficacy, Safety, and Tolerability of SAR440340/REGN3500/Itepekimab in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: AERIFY-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC16750; U1111-1250-2787 (Registry Identifier: ICTRP); 2024-512013-41 (Registry Identifier: CTIS); 2020-001818-38 (EudraCT Number)
Record Dates: First submitted 2020-12-30; First posted 2021-01-08 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Itepekimab Q2W (Experimental): Subcutaneous (SC) administration of Itepekimab every 2 weeks (Q2W) for up to 52 weeks
  Interventions: Drug: Itepekimab SAR440340
- Itepekimab Q4W (Experimental): SC administration of Itepekimab every 4 weeks (Q4W) for up to 52 weeks, with alternating SC administration of matching placebo at the 2-week interval between active IMP
  Interventions: Drug: Itepekimab SAR440340; Drug: Placebo
- Placebo (Placebo Comparator): SC administration of matching placebo Q2W for up to 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itepekimab SAR440340 — Pharmaceutical form: solution for injection in pre-filled syringe Route of administration: subcutaneous
  Other Names: REGN3500
  Arms: Itepekimab Q2W; Itepekimab Q4W
Drug: Placebo — Pharmaceutical form: solution for injection in pre-filled syringe Route of administration: subcutaneous
  Arms: Itepekimab Q4W; Placebo

SUMMARY:
Primary Objective:

Evaluate the efficacy of itepekimab compared with placebo on the annualized rate of acute moderate-or-severe COPD exacerbations in former smokers with moderate-to-severe COPD

Secondary Objectives:

* Evaluate the efficacy of itepekimab compared with placebo on pulmonary function in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on occurrence of acute exacerbation of COPD (AECOPD) in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on severe AECOPD in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on corticosteroid-treated AECOPD in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on respiratory symptoms in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on Forced Expiratory Volume in 1 second (FEV1) slope in former smokers with moderate-to-severe COPD
* Evaluate the efficacy of itepekimab compared with placebo on health-related quality of life (HRQoL) as assessed by St. George's Respiratory Questionnaire (SGRQ) in former smokers with moderate-to-severe COPD
* Evaluate the safety and tolerability of itepekimab in former smokers with moderate-to-severe COPD
* Evaluate the pharmacokinetic (PK) profile of itepekimab in former smokers with moderate-to-severe COPD
* Evaluate immunogenicity to itepekimab in former smokers with moderate-to-severe COPD

DETAILED DESCRIPTION:
The study duration per participant:

* Screening period is 3-5 weeks
* Placebo-controlled treatment period is 52 weeks for first approximately 960 randomized participants, and 24 to 52 weeks for potential additional randomized participants
* Post-investigational medicinal product (IMP) treatment follow-up period is 20 weeks for participants not transitioning to the extension study LTS18133 Note: A long-term, double-blinded extension study (LTS18133) will be implemented to allow participants in this study to continue receiving active IMP for an additional period. Only participants completing their End-of-Treatment (EOT) visit per this study protocol will be offered to participate in the LTS18133 study.

ELIGIBILITY:
Inclusion criteria :

* Participant must be 40 to 85 years of age inclusive.
* Physician diagnosis of COPD for at least 1 year (based on Global Initiative for Chronic Obstructive Lung Disease [GOLD] definition).
* Smoking history of ≥10 pack-years, but who are not currently smoking, and smoking cessation must have occurred ≥6 months prior to Screening (Visit 1A) with an intention to quit permanently.
* Participants with moderate-to-severe COPD
* Participant-reported history of signs and symptoms of chronic bronchitis (chronic productive cough for at least 3 months in the year prior to screening in a participant in whom other causes of chronic cough [eg, inadequately treated gastroesophageal reflux or chronic rhinosinusitis; or clinical diagnosis of bronchiectasis] has been excluded).
* Documented history of high exacerbation risk defined as having had ≥2 moderate or ≥1 severe exacerbations within the year prior to Screening (Visit 1A), with at least 1 exacerbation treated with systemic corticosteroids. At least one exacerbation must have occurred while participants were on their current controller therapy:

  * Moderate exacerbations will be recorded by the Investigator and are defined as acute worsening of respiratory symptoms that requires either systemic corticosteroids (IM, IV, or oral) and/or antibiotics.
  * Severe exacerbations will be recorded by the Investigator and are defined as AECOPD that require hospitalization or observation for >24 hours in emergency department/urgent care facility.
* Participants with standard of care controller therapy, for ≥3 months prior to Screening (Visit 1A) and at a stable dose of controller therapy for at least 1 month prior to the screening, including either: inhaled corticosteroid (ICS) + long-acting beta-agonist (LABA), long-acting muscarinic antagonist (LAMA) + LABA or LAMA + LABA + ICS.
* Body mass index (BMI) ≥18.0 kg/m^2, or BMI ≥16.0 kg/m^2 for participants enrolled in East-Asian countries.
* Female participant is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * not a women of child-bearing potential (WOCBP) OR
  * a WOCBP who agrees to follow the contraceptive guidance during the intervention period and for at least 20 weeks after the last dose of study intervention.

Exclusion criteria:

* Current diagnosis of asthma according to the Global Initiative for Asthma (GINA) guidelines, or documented history of asthma unless asthma resolved before 18 years of age and has not recurred.
* Active smoking or vaping of any products (eg, nicotine, tetrahydrocannabinol [THC]) within 6 months prior to Screening (Visit 1A).
* Clinically significant new abnormal electrocardiogram (ECG) within 6 months prior to, or at Screening (Visit 1A) that may affect the participant's participation in the study.
* Clinically significant and current pulmonary disease other than COPD, eg, sarcoidosis, interstitial lung disease, bronchiectasis (clinical diagnosis), diagnosis of α-1 anti-trypsin deficiency, or another diagnosed pulmonary disease.
* Diagnosis of cor pulmonale, evidence of right cardiac failure, or moderate-to-severe pulmonary hypertension.
* Hypercapnia requiring bilevel positive airway pressure (BiPAP).
* Moderate or severe exacerbation of COPD (AECOPD) within 4 weeks prior to Screening (Visit 1A).
* Prior history of / planned: lung pneumonectomy for any reason, or lung volume reduction procedures (including bronchoscopic volume reduction) for COPD. Note: Surgical biopsy, or segmentectomy, or wedge resection, or lobectomy for other diseases would not be excluded.
* Unstable ischemic heart disease, including acute myocardial infarction within the past 1 year prior to Screening, or unstable angina in the 6 months prior to Screening (Visit 1A).
* Cardiac arrhythmias including paroxysmal (eg, intermittent) atrial fibrillation.
* Uncontrolled hypertension (ie, systolic blood pressure [BP] >180 mm Hg or diastolic BP >110 mm Hg with or without use of anti-hypertensive therapy).
* Participants with active tuberculosis (TB), latent TB, a history of incompletely treated TB, suspected extrapulmonary TB infection (TBI), or who are at high risk of contracting TB (such as close contact with individuals with active or latent TB) or received Bacillus Calmette-Guérin (BCG)-vaccination within 12 weeks prior to Screening (Visit 1A).
* History of human immunodeficiency virus (HIV) infection or positive HIV 1/2 serology at Screening (Visit 1A).
* Suspicion of, or confirmed, coronavirus disease 2019 (COVID-19) infection or in contact with known exposure to COVID-19 at Screening (Visit 1A); known history of COVID-19 infection within 4 weeks prior to Screening (Visit 1A); history of requiring mechanical ventilation or extracorporeal membrane oxygenation (ECMO) secondary to COVID-19 within 3 months prior to sScreening (Visit 1A); participants who have had a COVID-19 infection prior Screening (Visit 1A) who have not yet sufficiently recovered to participate in the procedures of a clinical trial.
* Evidence of acute or chronic infection requiring systemic treatment with antibacterial, antiviral, antifungal, antiparasitic, or antiprotozoal medications within 4 weeks before Screening (Visit 1A), significant viral infections within 4 weeks before Screening (Visit 1A) that may not have been treated with antiviral treatment (eg, influenza receiving only symptomatic treatment).
* Participants with active autoimmune disease or participants using immunosuppressive therapy for autoimmune disease (eg, rheumatoid arthritis, inflammatory bowel disease, primary biliary cirrhosis, systemic lupus erythematosus, multiple sclerosis.
* History of malignancy within 5 years before Screening (Visit 1A), except completely treated in situ carcinoma of the cervix, completely treated and resolved nonmetastatic squamous or basal cell carcinoma of the skin.
* Previous use of itepekimab.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1127 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Annualized rate of moderate or severe acute exacerbation of COPD (AECOPD) | Baseline up to End Of Treatment (EOT) (Week 52 for initial randomized participants, Week 24 to 52 for potential additional randomized participants)
  Annualized rate of moderate or severe AECOPD over the placebo-controlled treatment period

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) | Baseline to Week 24
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Change from baseline in post-BD FEV1 | Baseline to Week 24 and Week 52
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Change from baseline in pre-BD FEV1 | Baseline to Week 52
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Time to first moderate or severe AECOPD | Baseline through EOT (Week 52 for initial randomized participants, Week 24 to 52 for potential additional randomized participants)
  Time to first moderate or severe AECOPD over the placebo-controlled treatment period
Annualized rate of severe AECOPD | Baseline up to EOT (Week 52 for initial randomized participants, Week 24 to 52 for potential additional randomized participants)
  Annualized rate of severe AECOPD over the placebo-controlled treatment period
Time to first severe AECOPD | Baseline through EOT (Week 52 for initial randomized participants, Week 24 to 52 for potential additional randomized participants)
  Time to first severe AECOPD over the placebo-controlled treatment period.
Annualized rate of corticosteroid-treated AECOPD | Baseline up to EOT (Week 52 for initial randomized participants, Week 24 to 52 for potential additional randomized participants)
  Annualized rate of corticosteroid-treated AECOPD over the placebo-controlled treatment period.
Change from baseline in Evaluating Respiratory Symptoms in COPD (E-RS:COPD) total score | Baseline to Week 24 and Week 52
  The E-RS: COPD is administered as a part of the 14-item EXACT questionnaire and is completed on a daily basis.The 11-item E-RS:COPD assesses severity of respiratory symptoms overall and severity of individual symptoms such as breathlessness, cough and sputum, and chest symptoms The total score of E-RS:COPD ranges from 0 to 40, with higher values indicating more severe respiratory symptoms.
Rate of change in post-BD FEV1 (L) from baseline (post-BD FEV1 slope) | Baseline up to EOT (Week 52 for initial randomized participants, Week 24 to 52 for potential additional randomized participants)
  FEV1 is the volume of air exhaled in the first second of a forced expiration as measured by spirometer.
Change from baseline in St. George''s Respiratory Questionnaire (SGRQ) total score | Baseline to Week 24 and Week 52
  The SGRQ is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation. A global score ranges from 0 to 100. Scores by dimension are calculated for 3 domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A lower score indicates better quality of life.
Proportion of participants with a decrease from baseline of at least 4 points in SGRQ total score | Baseline to Week 24 and Week 52
  The SGRQ is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation. A global score ranges from 0 to 100. Scores by dimension are calculated for 3 domains: Symptoms, Activity and Impacts (Psycho-social) as well as a total score. A lower score indicates better quality of life.
Incidence of treatment-emergent adverse events (TEAEs), adverse event of special interests (AESIs), serious adverse events (SAEs), and adverse events (AEs) leading to permanent treatment discontinuation | Baseline up to End-of-Study (EOS) (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)
Incidence of potentially clinically significant laboratory test, vital signs, and electrocardiogram (ECGs) abnormalities | Baseline up to EOS (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)
Functional itepekimab concentrations in serum | Baseline up to EOS (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)
Incidence of treatment-emergent anti-itepekimab antibodies responses | Baseline up to EOS (Up to Week 72 for participants not transitioning to the extension study LTS18133; Up to Week 52 for participants transitioning to the extension study LTS18133)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (248):
- United States (86):
  - University of Alabama at Birmingham Site Number : 8400012, Birmingham, Alabama
  - Jasper Summit Research Site Number : 8400178, Jasper, Alabama
  - Chandler Clinical Trials (Elite Clinical Network) Site Number : 8400034, Chandler, Arizona
  - Pulmonary Associates Site Number : 8400392, Phoenix, Arizona
  - Noble Clinical Research Site Number : 8400182, Tucson, Arizona
  - Tucson Clinical Research Institute Site Number : 8400431, Tucson, Arizona
  - California Research Institute Site Number : 8400400, Huntington Park, California
  - Modena Allergy + Asthma Site Number : 8400036, La Jolla, California
  - Imax Clinical Trials LLC 1 Site Number : 8400419, La Palma, California
  - Downtown LA Research Center Inc. Site Number : 8400027, Los Angeles, California
  - MACRO Trials Site Number : 8400030, Los Angeles, California
  - Antelope Valley Clinical Trials Site Number : 8400003, Northridge, California
  - ~Alpine Clinical Research Center Site Number : 8400180, Boulder, Colorado
  - Innovative Clinical Research Site Number : 8400017, Lafayette, Colorado
  - Clin Research W Florida Site Number : 8400004, Clearwater, Florida
  - Beautiful Minds Clinical Research Center Site Number : 8400037, Cutler Bay, Florida
  - Indago Research and Health Center Site Number : 8400187, Hialeah, Florida
  - Advanced Clinical Research Site Number : 8400409, Kendall, Florida
  - Advanced Pulmonary Research Institute Site Number : 8400455, Loxahatchee Groves, Florida
  - University of Miami/Miami VA Medical Center Site Number : 8400026, Miami, Florida
  - DL Research Solutions Inc Site Number : 8400033, Miami, Florida
  - My Community Research Center Site Number : 8400347, Miami, Florida
  - Reliant Medical Research Site Number : 8400397, Miami, Florida
  - Research Institute of South Florida,Inc Site Number : 8400006, Miami, Florida
  - PROLIVE MEDICAL RESEARCH Site Number : 8400420, Miami, Florida
  - Reed Medical Research Site Number : 8400032, Miami, Florida
  - High Quality Research Site Number : 8400406, Miami, Florida
  - Deluxe Health Center Site Number : 8400188, Miami Lakes, Florida
  - Florida Institute for Clinical Research Site Number : 8400013, Orlando, Florida
  - Tellabio International Research Services Site Number : 8400411, Pembroke Pines, Florida
  - Avanza Medical Research Center Site Number : 8400376, Pensacola, Florida
  - Broward Pulmonary and Sleep Specialists Site Number : 8400031, Plantation, Florida
  - Coastal Medical Research Institute Site Number : 8400044, St. Petersburg, Florida
  - Pasadena Center for Medical Research Site Number : 8400043, St. Petersburg, Florida
  - AdtreMed Site Number : 8400442, Tampa, Florida
  - Premier Medical Associates Site Number : 8400388, The Villages, Florida
  - Appalachian Clinical Research Site Number : 8400024, Adairsville, Georgia
  - Covenant Pulmonary Critical Care Site Number : 8400183, Atlanta, Georgia
  - David Kavtaradze MD, Inc. Site Number : 8400029, Cordele, Georgia
  - Alpha Clinical Research Georgia Site Number : 8400190, Dunwoody, Georgia
  - Gwinnett Biomedical Research Site Number : 8400007, Lawrenceville, Georgia
  - GenHarp Clinical Solutions Site Number : 8400028, Evergreen Park, Illinois
  - ASHA Clinical Research Site Number : 8400408, Hammond, Indiana
  - Benchmark Research Site Number : 8400193, Covington, Louisiana
  - Paul Shapero, PC Site Number : 8400016, Bangor, Maine
  - Care Access Site Number : 8400276, Boston, Massachusetts
  - Care Access Site Number : 8400277, Boston, Massachusetts
  - Care Access Site Number : 8400278, Boston, Massachusetts
  - Care Access Site Number : 8400280, Boston, Massachusetts
  - Care Access Site Number : 8400281, Boston, Massachusetts
  - Exordia Medical Research, Inc. Site Number : 8400041, Fall River, Massachusetts
  - Revival Research Institute, LLC Site Number : 8400191, Dearborn, Michigan
  - Advanced Pulmonary Research Institute of Michigan Site Number : 8400403, Warren, Michigan
  - Hannibal Clinic Site Number : 8400383, Hannibal, Missouri
  - Midwest Chest Consultants, P.C. Site Number : 8400002, Saint Charles, Missouri
  - Hendeson Clinical Trials Site Number : 8400365, Henderson, Nevada
  - Northwell Health Site Number : 8400019, Mount Kisco, New York
  - WellNow Urgent Care and Clinical Research Site Number : 8400378, Schenectady, New York
  - Gastonia Pharmaceutical Research Site Number : 8400010, Gastonia, North Carolina
  - East Carolina University Brody School Of Medicine Site Number : 8400022, Greenville, North Carolina
  - Carolina Research Center Site Number : 8400005, Shelby, North Carolina
  - Accellacare Site Number : 8400001, Wilmington, North Carolina
  - Southeastern Research Center Site Number : 8400011, Winston-Salem, North Carolina
  - Bernstein Clinical Research Center Site Number : 8400014, Cincinnati, Ohio
  - WellNow Urgent Care and Research Site Number : 8400039, Springdale, Ohio
  - Clinical Research of Central PA Site Number : 8400023, DuBois, Pennsylvania
  - Bogan Sleep Consultants Site Number : 8400181, Columbia, South Carolina
  - Clinical Research of Rock Hill Site Number : 8400008, Rock Hill, South Carolina
  - REX Clinical Trials Site Number : 8400371, Beaumont, Texas
  - Clinrx Research Site Number : 8400021, Carrollton, Texas
  - Austin Pulmonary Consultants Site Number : 8400035, Cedar Park, Texas
  - Corsicana Medical Research, LLC Site Number : 8400018, Corsicana, Texas
  - Premier Pulmonary Critical Care and Sleep Medicine Site Number : 8400440, Denison, Texas
  - Texas Tech University Health Sciences Center Site Number : 8400189, El Paso, Texas
  - The Methodist Hospital Research Institute Site Number : 8400194, Houston, Texas
  - Biopharma Informatic - Cardiff Avenue - PPDS Site Number : 8400038, Houston, Texas
  - Santa Clara Family Clinic Site Number : 8400398, Houston, Texas
  - Metroplex Pulmonary and Sleep Center Site Number : 8400015, McKinney, Texas
  - PRX Research Site Number : 8400380, Mesquite, Texas
  - The Lung and Sleep Research Institute of North Texas Site Number : 8400417, North Richland Hills, Texas
  - Clincove: Plano Primary Care Clinic Site Number : 8400424, Plano, Texas
  - EPW Curesearch Dallas (Advanced Family Medical Care) Site Number : 8400414, Plano, Texas
  - Advance Lung and Sleep Center Site Number : 8400040, Sherman, Texas
  - Sherman Clinical Research Site Number : 8400009, Sherman, Texas
  - DM Clinical Research Site Number : 8400179, Tomball, Texas
  - Clearlake Specialties Site Number : 8400025, Webster, Texas
- Argentina (5):
  - Investigational Site Number : 0320001, CABA, Buenos Aires
  - Investigational Site Number : 0320002, CABA, Buenos Aires
  - Investigational Site Number : 0320005, La Plata, Buenos Aires
  - Investigational Site Number : 0320003, Rosario, Santa Fe Province
  - Investigational Site Number : 0320004, Mendoza
- Bulgaria (9):
  - Investigational Site Number : 1000005, Dimitrovgrad
  - Investigational Site Number : 1000001, Sofia
  - Investigational Site Number : 1000004, Sofia
  - Investigational Site Number : 1000002, Sofia
  - Investigational Site Number : 1000009, Sofia
  - Investigational Site Number : 1000006, Stara Zagora
  - Investigational Site Number : 1000003, Stara Zagora
  - Investigational Site Number : 1000007, Veliko Tyrnovo
  - Investigational Site Number : 1000008, Vidin
- Chile (9):
  - Investigational Site Number : 1520008, Temuco, La Araucanía
  - Investigational Site Number : 1520007, Curicó, Maule Region
  - Investigational Site Number : 1520002, Talca, Maule Region
  - Investigational Site Number : 1520009, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520005, Quillota, Región de Valparaíso
- China (42):
  - Investigational Site Number : 1560003, Baotou
  - Investigational Site Number : 1560004, Beijing
  - Investigational Site Number : 1560030, Beijing
  - Investigational Site Number : 1560014, Beijing
  - Investigational Site Number : 1560002, Changchun
  - Investigational Site Number : 1560012, Changsha
  - Investigational Site Number : 1560013, Changsha
  - Investigational Site Number : 1560047, Changsha
  - Investigational Site Number : 1560001, Chengdu
  - Investigational Site Number : 1560040, Chengdu
  - Investigational Site Number : 1560032, Chongqing
  - Investigational Site Number : 1560006, Guangzhou
  - Investigational Site Number : 1560025, Guangzhou
  - Investigational Site Number : 1560036, Haikou
  - Investigational Site Number : 1560022, Hangzhou
  - Investigational Site Number : 1560039, Hangzhou
  - Investigational Site Number : 1560017, Hefei
  - Investigational Site Number : 1560008, Hohhot
  - Investigational Site Number : 1560010, Hohhot
  - Investigational Site Number : 1560044, Jinan
  - Investigational Site Number : 1560027, Jinan
  - Investigational Site Number : 1560031, Nanchang
  - Investigational Site Number : 1560035, Nanjing
  - Investigational Site Number : 1560023, Nanning
  - Investigational Site Number : 1560015, Pingxiang
  - Investigational Site Number : 1560043, Shanghai
  - Investigational Site Number : 1560034, Shanghai
  - Investigational Site Number : 1560009, Shanghai
  - Investigational Site Number : 1560045, Shanghai
  - Investigational Site Number : 1560005, Shenyang
  - Investigational Site Number : 1560020, Shenzhen
  - Investigational Site Number : 1560028, Shijiazhuang
  - Investigational Site Number : 1560024, Tianjin
  - Investigational Site Number : 1560019, Wenzhou
  - Investigational Site Number : 1560029, Wuhan
  - Investigational Site Number : 1560016, Xi'an
  - Investigational Site Number : 1560046, Xiangtan
  - Investigational Site Number : 1560007, Xuzhou
  - Investigational Site Number : 1560026, Yangzhou
  - Investigational Site Number : 1560041, Zhanjiang
  - Investigational Site Number : 1560042, Zhengzhou
  - Investigational Site Number : 1560048, Zhongshan
- Czechia (6):
  - Investigational Site Number : 2030006, Havlíčkův Brod
  - Investigational Site Number : 2030001, Jindrichuv Hradec III
  - Investigational Site Number : 2030004, Ostrava
  - Investigational Site Number : 2030002, Prague
  - Investigational Site Number : 2030003, Prague
  - Investigational Site Number : 2030005, Praha 5 - Radotin
- Georgia (3):
  - Investigational Site Number : 2680002, Tbilisi
  - Investigational Site Number : 2680003, Tbilisi
  - Investigational Site Number : 2680001, Tbilisi
- Greece (7):
  - Investigational Site Number : 3000005, Athens
  - Investigational Site Number : 3000006, Athens
  - Investigational Site Number : 3000004, Heraklion
  - Investigational Site Number : 3000001, Ioannina
  - Investigational Site Number : 3000007, Larissa
  - Investigational Site Number : 3000008, Palaio Faliro, Athens
  - Investigational Site Number : 3000002, Thessaloniki
- Hungary (4):
  - Investigational Site Number : 3480004, Debrecen
  - Investigational Site Number : 3480001, Gödöllö
  - Investigational Site Number : 3480002, Mosonmagyaróvár
  - Investigational Site Number : 3480003, Pécs
- India (6):
  - Investigational Site Number : 3560002, Coimbatore
  - Investigational Site Number : 3560005, Hyderabad
  - Investigational Site Number : 3560004, Jaipur
  - Investigational Site Number : 3560001, Kozhikode
  - Investigational Site Number : 3560007, Mumbai
  - Investigational Site Number : 3560003, Nagpur
- Israel (8):
  - Investigational Site Number : 3760008, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760002, Jerusalem
  - Investigational Site Number : 3760006, Kfar Saba
  - Investigational Site Number : 3760001, Petah Tikva
  - Investigational Site Number : 3760009, Ramat Gan
  - Investigational Site Number : 3760004, Rehovot
  - Investigational Site Number : 3760007, Tel Aviv
- Italy (5):
  - Investigational Site Number : 3800004, Foggia, Apulia
  - Investigational Site Number : 3800003, Rozzano, Milano
  - Investigational Site Number : 3800005, Catania
  - Investigational Site Number : 3800001, Ferrara
  - Investigational Site Number : 3800007, Verona
- Investigational Site Number : 4800001, Quatre Bornes, Mauritius
- Mexico (10):
  - Investigational Site Number : 4840001, Guadalajara, Jalisco
  - Investigational Site Number : 4840011, Guadalajara, Jalisco
  - Investigational Site Number : 4840010, Guadalajara, Jalisco
  - Investigational Site Number : 4840002, Mexico City, Mexico City
  - Investigational Site Number : 4840007, Cuernavaca, Morelos
  - Investigational Site Number : 4840016, Oaxaca City, Oaxaca
  - Investigational Site Number : 4840003, San Juan del Río, Querétaro
  - Investigational Site Number : 4840013, Aguascalientes
  - Investigational Site Number : 4840004, Benito Juárez
  - Investigational Site Number : 4840014, Oaxaca City
- Poland (4):
  - Investigational Site Number : 6160004, Wroclaw, Lower Silesian Voivodeship
  - Investigational Site Number : 6160003, Warsaw, Masovian Voivodeship
  - Investigational Site Number : 6160001, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160002, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Romania (9):
  - Investigational Site Number : 6420005, Bragadiru
  - Investigational Site Number : 6420006, Brasov
  - Investigational Site Number : 6420012, Bucaresti
  - Investigational Site Number : 6420002, Cluj-Napoca
  - Investigational Site Number : 6420007, Codlea
  - Investigational Site Number : 6420010, Deva
  - Investigational Site Number : 6420001, Iași
  - Investigational Site Number : 6420009, Oradea
  - Investigational Site Number : 6420003, Timișoara
- Russia (5):
  - Investigational Site Number : 6430001, Moscow
  - Investigational Site Number : 6430003, Moscow
  - Investigational Site Number : 6430002, Moscow
  - Investigational Site Number : 6430005, Saint Petersburg
  - Investigational Site Number : 6430006, Saint Petersburg
- Slovakia (7):
  - Investigational Site Number : 7030009, Bardejov
  - Investigational Site Number : 7030007, Humenné
  - Investigational Site Number : 7030003, Levice
  - Investigational Site Number : 7030011, Martin
  - Investigational Site Number : 7030002, Poprad
  - Investigational Site Number : 7030010, Prešov
  - Investigational Site Number : 7030001, Spišská Nová Ves
- Taiwan (6):
  - Investigational Site Number : 1580005, Kaohsiung City
  - Investigational Site Number : 1580002, New Taipei City
  - Investigational Site Number : 1580006, Taichung
  - Investigational Site Number : 1580004, Taipei
  - Investigational Site Number : 1580003, Taipei
  - Investigational Site Number : 1580008, Yunlin
- Ukraine (8):
  - Investigational Site Number : 8040003, Ivano-Frankivsk
  - Investigational Site Number : 8040007, Ivano-Frankivsk
  - Investigational Site Number : 8040008, Kharkiv
  - Investigational Site Number : 8040006, Kharkiv
  - Investigational Site Number : 8040004, Kyiv
  - Investigational Site Number : 8040001, Kyiv
  - Investigational Site Number : 8040005, Kyiv
  - Investigational Site Number : 8040011, Kyiv
- United Kingdom (8):
  - Investigational Site Number : 8260004, Portsmouth, Hampshire
  - Investigational Site Number : 8260015, Ashton-under-Lyne, Lancashire
  - Investigational Site Number : 8260010, Wigan, Lancashire
  - Investigational Site Number : 8260016, Salford, Manchester
  - Investigational Site Number : 8260003, Bradford
  - Investigational Site Number : 8260014, Heston
  - Investigational Site Number : 8260001, London
  - Investigational Site Number : 8260013, Redruth

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC16750 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25254&tenant=MT_SNY_9011